CLINICAL TRIAL: NCT00487916
Title: Phase 1 Study of the Safety, Reactogenicity and Immunogenicity of AMA1-C1/ISA 720: A Blood Stage Vaccine for Plasmodium Falciparum
Brief Title: Phase 1 Study of the Safety, Reactogenicity, and Immunogenicity of AMA1-C1/ISA 720: Blood Stage Vaccine for Plasmodium Falciparum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 999907170; 07-I-N170
Record Dates: First submitted 2007-06-16; First posted 2007-06-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-22

CONDITIONS: Malaria
Keywords: Blood Stage; Investigational; Vaccine; Malaria; Healthy Volunteer; HV
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Drug: AMA1-C1/ISA 720

SUMMARY:
This study will evaluate the safety and effectiveness of a vaccine called AMA1-C1/ISA. Malaria is a serious infection of red blood cells caused by a parasite. There are 300 to 500 million malaria cases worldwide each year. About 2 to 3 million deaths annually are from malaria alone or along with other diseases. Researchers hope to find a vaccine to fight malaria.

Patients ages 18 to 45 who are in good health, are not pregnant or breast feeding, have no history of malaria, and have not lived for more than 1 month in an area where malaria is prevalent may be eligible for this study. There will be 28 participants, each assigned to one of three dose groups: 12 get 5 microg, 12 get 20 microg, and 4 get 80 microg of AMA 1-C1 formulated in ISA 720. The vaccine might block the parasite from entering red blood cells and causing disease. This study is the first time the vaccine will be given to human beings for testing.

Patients will have a medical history, physical exam, laboratory tests, and pregnancy tests. The study will last 48 weeks. One or two vaccinations are given by injection, at least 12 weeks apart. After each vaccination, patients will be asked to stay in the clinic for at least 30 minutes for observation. They will return to the clinic on Days 1, 3, 7, 14, 28, and 56 after each vaccination. There will be a check of vital signs, brief physical exam, history of symptoms and medications taken since the last visit, and blood tests to check for vaccine safety and effectiveness. Photographs of the injection site on the arm may be taken. Patients will receive a thermometer, diary card, and plastic measuring device. Each day they will record their temperatures and any symptoms, and measure the size of any reactions at the vaccination site. They will be asked to do this for 27 days after vaccinations.

After injections, there may be pain, swelling, and redness at the vaccination site, and limitation of arm movement. General side effects from the vaccine may be fever, chills, headache, fatigue, and muscle and joint pain. Patients will be asked if they agree to have researchers keep any unused serum samples, for use only in research into malaria and other diseases. Genetic testing would not be done on those samples. Stored samples will be labeled with a code, and information is kept private.

DETAILED DESCRIPTION:
AMA1-C1 with Montanide ISA 720, is a blood stage malaria vaccine candidate. The objectives of this phase 1 trial are to study the safety, reactogenicity, and immunogenicity of this vaccine and to assess the level, kinetics, and the in vitro biological activity of the antibody response it induces. The study is an open label, dose escalation, phase 1 clinical trial in healthy adult volunteers. Volunteers will be screened and 28 participants will be enrolled into 3 dose cohorts. Cohort 1 will receive 5 micrograms of AMA1-C1/ISA 720 at each injection, Cohort 2 will receive 20 micrograms, and Cohort 3 will receive 80 micrograms. Cohorts 1 and 2 will receive 2 injections, 3 months apart. Cohort 3 will receive only 1 vaccination. Safety outcome measures are local and systemic (including laboratory) adverse events. Immune responses to vaccination will be measured by enzyme-linked immunosorbent assay (ELISA) and parasite growth inhibition assay (GIA), and will be compared among dose groups.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males or females between 18 and 45 years, inclusive.
  2. Good general health as determined by means of the screening procedure.
  3. Available for the duration of the trial (48 weeks).
  4. Willingness to participate in the study as evidenced by signing the informed consent document.
  5. For female subjects: Negative pregnancy tests at Screening and Day 0, in conjunction with a history indicating a low probability of pregnancy in the opinion of the physician. Sexually active females of childbearing potential will be required to be correctly using an efficacious method of contraception for at least 1 month before randomization and during the on-study phase to Month 7. Female subjects unable to become pregnant must have this documented (e.g. tubal ligation, hysterectomy, or postmenopausal [at least one year since last menstrual period]).

EXCLUSION CRITERIA:

1. History of malaria, residence for more than 1 month in a malaria endemic area (as determined by interview), or plans to visit a malaria endemic area during the study period.
2. For female subjects: Positive pregnancy test at screening or Day 0, as well as those currently lactating and breast feeding.
3. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, chronic infectious or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
4. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.
5. Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25 times the upper limit of normal of the testing laboratory).
6. Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory, or more than trace protein or blood on urine dipstick testing confirmed by repeat testing of clean-catch, midstream sample). (More than trace blood on urine dipstick will not exclude a female who is actively menstruating).
7. Laboratory evidence of hematologic disease (absolute leukocyte count less than 3000/mm(3) or greater than 11,500/mm(3); hemoglobin less than 0.9 times the lower limit of normal of the testing laboratory, by gender; absolute granulocyte count less than 1300/mm(3); absolute lymphocyte count less than 1000/mm(3); or platelet count less than 11,000/mm(3)).
8. Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
9. Participation in another investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing.
10. Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
11. History of a severe allergic reaction or anaphylaxis.
12. Severe asthma. This will be defined as:

    * Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or parenteral corticosteroids.
    * Clinically significant reactive airway disease that does not respond to bronchodilators.
13. Positive ELISA for anti-HCV.
14. Positive hepatitis B surface antigen (HBsAg) by ELISA.
15. Positive ELISA for anti-HIV.
16. Use of systemic corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.
17. Receipt of a live vaccine within past 4 weeks or non-live vaccine within past 2 weeks prior to entry into the study.
18. History of a surgical splenectomy.
19. Receipt of blood products within the past 6 months.
20. Previous receipt of an investigational malaria vaccine.
21. History of a known allergy to nickel.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150
Dates: Start 2007-06-13; Primary Completion 2009-02-05 (Actual); Study Completion 2009-02-05 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and reactogenicity of the AMA1-C1/ISA 720 vaccine; and to determine the frequency of systemic and local AEs as recorded for 28 days following each vaccination.

SECONDARY OUTCOMES:
Assessment of the level, kinetics and the in-vitro biological activity of the antibody response to AMA1-FVO and AMA1-3D7.

CONTACTS AND LOCATIONS:
Locations (1):
- QIMR - CLive Berghofer Cancer Research Centre, Herston, Australia

REFERENCES:
- [Background] Narum DL, Thomas AW. Differential localization of full-length and processed forms of PF83/AMA-1 an apical membrane antigen of Plasmodium falciparum merozoites. Mol Biochem Parasitol. 1994 Sep;67(1):59-68. doi: 10.1016/0166-6851(94)90096-5. PMID 7838184
- [Background] Crewther PE, Culvenor JG, Silva A, Cooper JA, Anders RF. Plasmodium falciparum: two antigens of similar size are located in different compartments of the rhoptry. Exp Parasitol. 1990 Feb;70(2):193-206. doi: 10.1016/0014-4894(90)90100-q. PMID 2404781
- [Background] Waters AP, Thomas AW, Deans JA, Mitchell GH, Hudson DE, Miller LH, McCutchan TF, Cohen S. A merozoite receptor protein from Plasmodium knowlesi is highly conserved and distributed throughout Plasmodium. J Biol Chem. 1990 Oct 15;265(29):17974-9. PMID 2211675